CLINICAL TRIAL: NCT07113951
Title: Diagnostic Application of Microbiological Fluorescence Rapid On-site Evaluation Combined With Artificial Intelligence in Severe Pneumonia: a Multi-center Prospective Study
Brief Title: Diagnostic Application of AI-ROSE in Severe Pneumonia
Status: Enrolling by invitation | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-SR-567
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Severe Pneumonia; Bacterial Infections
Keywords: Severe Pneumonia; artificial intelligence; Rapid on-site evaluation; Diagnosis
MeSH Terms: conditions — Pneumonia; Bacterial Infections; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
AI-ROSE is an innovative immunofluorescence staining combined with artificial intelligence image analysis technology that uses a fully automated fluorescence microscope to image pathogens in real time. AI algorithms automatically identify pathogen types (such as bacteria, fungi, etc.) and cellular backgrounds, quickly interpret results, and automatically issue color graphic reports for clinical doctors to take earlier and more accurate targeted treatment for critically ill patients. This study used bronchoalveolar lavage fluid as a biological sample and compared it with traditional examination methods to analyze the diagnostic accuracy and clinical practicality of AI-ROSE in patients with severe pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* The preliminary clinical diagnosis is a patient with lower respiratory tract infection
* Meets the criteria for severe pneumonia, which means one of the following conditions exists: ① Main criteria: septic shock requiring vasoactive drug support; Respiratory failure requiring mechanical ventilation; ② Secondary criteria: Meet at least 3 or more criteria, including respiratory rate>30 times/minute; Oxygenation index (PaO ₂/FiO ₂)<250; Multiple leaf segment infiltration; Consciousness disorders/orientation disorders; Urea nitrogen level>20mg/dL; White blood cell count<4 * 10 ^ 9/L; platelet count<100 * 10 ^ 9/L; core body temperature<36.8 ° C; hypotension requiring active fluid resuscitation
* The patient agrees to undergo bronchoscopy and bronchoalveolar lavage, and agrees to perform AI-ROSE testing on the bronchoalveolar lavage fluid

Exclusion Criteria:

* Patients with poor basic condition, severe illness, and inability to tolerate bronchoscopy examination
* The bronchoalveolar lavage fluid sample is not qualified

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Infected severe pneumonia patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparing the diagnostic accuracy of AI-ROSE with traditional bronchoalveolar lavage fluid examination methods. | 2026-3-31

CONTACTS AND LOCATIONS:
Overall Officials: Wenkui Sun, Study Director — First Affiliated Hospital of Nanjing Medical University Nanjing
Locations (1):
- Fluorescence Biological Microscope, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No